CLINICAL TRIAL: NCT01990053
Title: Pilot Study Assessing Computerized Cognitive Behavioral Therapy for Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Daniel R. Strunk, Associate Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013B0307
Record Dates: First submitted 2013-10-28; First posted 2013-11-21 (Estimated); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Beating the Blues (Experimental): Beating the Blues plus helper support.
  Interventions: Behavioral: Beating the Blues
- Waitlist Condition (No Intervention): Eight week waitlist condition group parallel to the immediate treatment condition with optional entrance into the Beating the Blues after the first eight weeks

INTERVENTIONS:
Behavioral: Beating the Blues — The BtB program guides patients through a series of 8 fully automated online lessons intended to help them identify and change problematic patterns of thinking and behavior that maintain depression. Support will be provided by licensed professional therapists over the phone or via email.
  Other Names: Beating the Blues (BtB)
  Arms: Beating the Blues

SUMMARY:
Standard treatments for depression in specialty care settings are effective but resources for delivering empirically supported psychotherapies are often limited. Computerized cognitive behavioral therapy (cCBT) is an effective and highly scalable treatment for depression that might help expand services in psychiatric settings, however, little is known about its efficacy in this population. The present study aims to establish the efficacy of a internet-delivered cCBT program ("Beating the Blues") plus email and telephone support for depression in a psychiatric outpatient clinic setting. The secondary aim is to pilot an assessment procedure designed to identify moderators of treatment effectiveness.

DETAILED DESCRIPTION:
Currently, outpatient psychiatric settings are plagued by long wait times and are often unable to accommodate all individuals seeking services. Furthermore, a lack of trained therapists in these settings means that many treatment seekers do not have access to empirically supported psychotherapeutic treatments such as cognitive behavioral therapy. "Beating the Blues" (BtB) is a computerized, internet-delivered, cognitive behavioral treatment for depression. BtB is highly scalable and might enable a larger proportion of individuals to receive cognitive behavioral therapy in a psychiatric setting while also reducing therapist time. Although computerized CBT interventions have proven effective in primary care settings, there is no research demonstrating the effectiveness of cCBT in secondary care settings in the United States. Thus the primary goal of the proposed research is to test the efficacy of BtB in a specialty care sample.

Patients presenting to these settings tend to have more severe and complex psychopathology than those presenting to primary care. Although BtB is likely effective, computerized treatments do carry a higher risk of dropout and non-response. Therefore, reliable and valid predictors of response are needed to determine who is most likely to respond to the treatment, versus who is likely to fail or drop out. Thus the second aim of the current proposal is to pilot an assessment procedure containing a number of potential predictors of cCBT response and investigate these predictors for inclusion in a larger validation study.

The current trial is a pilot study with a randomized waitlist control design with optional delayed treatment for individuals randomized to the waitlist condition. For the first phase, the investigators will enroll 90 treatment-seeking adults 18 or older recruited from a pool of individuals seeking outpatient psychiatric services at a hospital clinic. Sixty (n=60) individuals will be assigned immediate treatment group with BtB plus telephone and email support, and n=30 to the waitlist/delayed BtB plus telephone and email support group. Efficacy will be assessed over 8 weeks using the Hamilton Rating Scale for Depression (pre to post treatment) and the PHQ9 (measured at weeks 1-8). There will also be a 1-year follow-up survey with biweekly symptom assessments throughout the year for treatment responders (weeks 9-61). Potential predictors of outcome include demographics, CBT skills, personality measures, cognitive functioning, measures of attitudes and beliefs, social functioning, psychiatric comorbidity and depression illness characteristics, and psychophysiological measures. A second phase will enroll sixty individuals (n=60), who will be assigned immediate treatment group in order to validate the predictive model constructed during Phase 1.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Major Depressive Disorder (MDD) according to Diagnostic and Statistical Manual Fourth Edition criteria
* Able and willing to give informed consent
* Have access to a computer with an internet connection at home

Exclusion Criteria:

* History of bipolar affective disorder or psychosis
* Current Axis I disorder other than MDD if it constitutes the predominate aspect of the clinical presentation and if it requires treatment other than that being offered
* History of substance dependence in the past six months
* Subnormal intellectual potential (IQ below 80)
* Clear indication of secondary gain (e.g., court ordered treatment or compensation issues)
* Current suicide risk or significant intentional self-harm in the last six months sufficient to preclude treatment on an outpatient basis
* Discharge within six moths from a higher level of care (inpatient, partial hospital, or intensive outpatient treatment)
* Currently undergoing outpatient psychotherapy
* Current antidepressant medication treatment if the individual has had a change in medication over the past month or is planning a change in medication during the duration of the study
* Inability to read and write English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2014-04-14 (Actual); Primary Completion 2016-05-03 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
Change in Hamilton Rating Scale for Depression (HRSD) from 0 to 8 weeks | week 0, week 8
  The 17-item HRSD, modified to assess atypical symptoms, is a standard interview-administered measure of depressive symptom severity. The HRSD will be administered by study personnel supervised by the Principal Investigator.

SECONDARY OUTCOMES:
Change in Patient Health Questionnaire-9 (PHQ9) over 8 weeks | weeks 0-8
  The PHQ9 is a 9-item self-report measure based on the diagnostic criteria for major depression from the Diagnostic and Statistical Manual Fourth Edition (DSM-IV).

OTHER OUTCOMES:
Change in Generalized Anxiety Disorder-7 (GAD7) over 8 weeks | weeks 0-8
  The GAD7 is a 7-item self-report measure based on the diagnostic criteria for generalized anxiety disorder from the DSM-IV.
Change in Depression Anxiety and Stress Scale-21 (DASS21) over 8 weeks | week 0, week 8
  The DASS21 is a 21-item self-report scale measuring symptoms of depression, anxiety, and stress.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel R Strunk, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States